CLINICAL TRIAL: NCT07354958
Title: Impact of Diabetes-Related Metabolic Derangements on Clinical Outcomes in Hospitalized Patients With Chronic Kidney Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Rashad, Resident in Internal Medicine department at sohage university, Sohag University
Other Study IDs: Soh-Med--25-12-5MS
Record Dates: First submitted 2025-12-25; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Chronic Kidney Disease Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1. Diabetic CKD (known diagnosis or on antidiabetic therapy prior to admission). 2. Non-diabetic CKD
  Interventions: Behavioral: Primary aim 1. To assess the frequency of diabetes mellitus among hospitalized CKD patients. 2. To evaluate the frequency and types of metabolic abnormalities (e.g., hypoglycemia, diabetic ketoacidosi

INTERVENTIONS:
Behavioral: Primary aim 1. To assess the frequency of diabetes mellitus among hospitalized CKD patients. 2. To evaluate the frequency and types of metabolic abnormalities (e.g., hypoglycemia, diabetic ketoacidosi — Primary aim
  1. To assess the frequency of diabetes mellitus among hospitalized CKD patients.
  2. To evaluate the frequency and types of metabolic abnormalities (e.g., hypoglycemia, diabetic ketoacidosis/ hyperosmolar states, metabolic acidosis, dyslipidemia, electrolyte imbalance) in diabetic CKD patients.
  Secondary aim
  1. To evaluate the association between diabetes and diabetes-related metabolic derangements in-hospital adverse outcomes (major cardiovascular events, ICU admission, length of stay, infection rate, need for dialysis and mortality) among hospitalized patients with CKD.

SUMMARY:
This observational study will collect clinical and laboratory information from hospitalized patients with chronic kidney disease to identify diabetes mellitus and selected metabolic findings during hospitalization

DETAILED DESCRIPTION:
Hospitalized adult patients with chronic kidney disease will be included in this observational study. Information routinely recorded during hospitalization will be collected. This information will include the presence of diabetes mellitus and laboratory values related to blood glucose levels, electrolyte levels, and acid base balance. No study related interventions will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Known chronic kidney disease, defined as baseline estimated glomerular filtration rate less than 60 milliliters per minute per 1.73 square meters for at least 3 months, or documented chronic kidney disease stage 3 to 5 by prior medical records
* Hospitalized for any medical reason
* Consent provided

Exclusion Criteria:

* Acute single episode of reversible acute kidney injury with previously normal renal function (no established chronic kidney disease)
* Admission for palliative care or expected survival less than 24 hours
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A) Inclusion criteria:
  * Age ≥18 years.
  * Known CKD (baseline eGFR <60 mL/min/1.73 m² for ≥3 months) OR documented CKD stage 3-5 by prior records.
  * Hospitalized for any medical reason.
  * Consent provided.
  B) Exclusion criteria:
  * Acute single episode of reversible AKI with previously normal renal function (no established CKD).
  * Admission for palliative care /expected survival <24 hours.
  * Pregnancy.
  C) Patient groups (for analysis):
  Diabetes status:
  * Diabetic CKD (known diagnosis or on antidiabetic therapy prior to admission).
  * Non-diabetic CKD.
  D) Subgroups / Diabetic patient group: Metabolic derangement categories
  1. Acute hyperglycemia
     * Diabetic ketoacidosis (DKA) /hyperosmolar hyperglycemic state (HHS)
     * Patients without DKA or HHS
  2. Hypoglycemia
     * Hypoglycemia: any blood glucose <70 mg/dL (and severe <40 mg/dL).
     * Without Hypoglycemia episodes
  3. Metabolic acidosis arterial or venous HCO₃- <20 mmol/L or pH <7.35 with anion gap >12 as appropriate.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
In-Hospital Mortality | From admission until hospital discharge, assessed over a 6-month study enrollment period.
  Patient death from any cause occurring during the hospitalization period
New Requirement for In-Hospital Renal Replacement Therapy | From admission until hospital discharge, assessed over a 6-month study enrollment period.
  Initiation of dialysis in a patient who was not receiving renal replacement therapy at the time of hospital admission
Incidence of a Major In-Hospital Cardiovascular Composite Event | From admission until hospital discharge, assessed over a 6-month study enrollment period.
  A composite outcome defined as the first occurrence of any of the following during the hospitalization: myocardial infarction, stroke, or new-onset heart failure requiring inotropic support or mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided